CLINICAL TRIAL: NCT03718728
Title: The Effect of a Group Intervention Program Based on Acceptance and Mindfulness on the Physical and Emotional Well-being of Overweight and Obese Individuals; Mind&Life Project
Brief Title: Effect of a Group Intervention Program Based on Acceptance and Mindfulness on the Physical and Emotional Well-being of Overweight and Obese Individuals
Acronym: Mind&Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Edurne Maiz Aldalur, PhD, Lecturer of School Psychology, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSI2017-88583-R
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Adults; Mindfulness; Acceptance; Emotional eating
MeSH Terms: conditions — Overweight; Obesity; Emotional Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): A personalized diet and physical exercise recommendations.
  Interventions: Behavioral: Standard
- Mind&Life (standard + intervention) group (Experimental): A personalized diet and physical exercise recommendations plus the acceptance and mindfulness-based group intervention program.
  Interventions: Behavioral: Mind&Life; Behavioral: Standard

INTERVENTIONS:
Behavioral: Mind&Life — Acceptance and mindfulness-based group intervention program.
  Arms: Mind&Life (standard + intervention) group
Behavioral: Standard — Personalized diet and physical exercise recommendations.

SUMMARY:
The objective of the present study is to evaluate the effect of a 20-week group intervention program based on acceptance and mindfulness in emotional eating, weight loss, physiological parameters and the level of physical exercise, as well as in the quality-of-life and weight self-stigma of overweight and obese people on the short- and medium-term.

Design, participants, and method: A randomized clinical trial comprising a total of 110 overweight or obese (BMI ≥ 25) participants that are receiving medical treatment at Primary Care Centers, 20-65 years, will be included and randomly assigned to standard program (N=55) or standard + intervention program (N=55). The standard program group will receive the treatment as usual (TAU) that comprises 5 sessions (on a monthly basis) that will include a personalized diet and physical exercise recommendations, while the standard + intervention program group will receive the same TAU plus the acceptance and mindfulness-based group intervention program.

At baseline prior to randomization, after the intervention, and seven months after the program has finished anthropometric and body composition data, biochemical data in blood, waist circumference, blood pressure, eating habits, level of physical exercise, general health, emotional eating, quality-of-life, weight self-stigma, experiential avoidance, self-compassion level and mindfulness abilities will be evaluated.

It is hypothesized that the integrated treatment of obesity implementing a group intervention program based on acceptance and mindfulness could help to reduce the emotional eating, enhance weight loss, improve physiological parameters, increase the level of physical exercise, improve the quality of life and reduce the weight self-stigma of overweight and obese individuals.

DETAILED DESCRIPTION:
The standard program group will receive the TAU that comprises 5 monthly sessions of 30 minutes that will include a personalized diet and physical exercise recommendations.

The standard + intervention program group will receive the same TAU plus the acceptance and mindfulness-based group intervention program. The first ten sessions will be held weekly and the last five, biweekly. The duration of sessions will be 2 hours and will include a mindfulness practice, the session content (i.e. control as the problem, willingness, etc.), followed by a mindful eating practice to train the ability to pay attention to food and eating physical sensations. Finally, the session content will be briefly revised and practices for the week will be established.

The following measurements will be evaluated at baseline prior to randomization, after the intervention, and seven months after the program has finished: anthropometric and body composition data, that is, weight and fat and muscle mass percentage (Bio-electrical Impedance Analysis, TANITA) and height (SECA 227); biochemical data in blood; waist circumference (Holtain inelastic tape); blood pressure; eating habits (24h recall and PREDIMED); level of physical exercise (IPAQ); general health (GHQ-28); emotional eating (DEBQ); quality-of-life (IWQOL-Lite); weight self-stigma (WSSQ); experiential avoidance (AAQ-II); self-compassion level (SCS) and mindfulness abilities (FFMQ).

ELIGIBILITY:
Inclusion Criteria:

* Adults with overweight or obesity (estimated by BMI ≥ 25 and classified by the International Obesity Task Force, IOTF);
* Have asked for enrollment in nutritional treatment for weight loss in primary care units from Donostia-San Sebastian;
* Willingness to participate in the study.

Exclusion Criteria:

* Diagnosed with eating disorders; such as, Binge Eating Disorder, Anorexia or Bulimia;
* Diagnosed with any psychiatric disorder or intellectual disability that doesn't allow to carry out the intervention;
* Not to know sufficiently the language the intervention is carried out.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-11-03 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in Body Mass Index (BMI) measured by Bio-electrical Impedance Analysis (TANITA) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in Body Mass Index (BMI - kg/m2) will be measured by Bio-electrical Impedance Analysis (TANITA).
Changes in eating habits estimated by 24h recall and PREDIMED questionnaire | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in eating habits will be estimated by 24h recall and PREDIMED questionnaire which is a questionnaire to assess the adherence to the Mediterranean diet, 0 being the minimum total score and 14 the maximum total score. Higher values represent a higher adherence to the Mediterranean diet.
Changes in the level of physical exercise estimated by the International Physical Activity Questionnaire (IPAQ) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in the level of physical exercise will be estimated by the International Physical Activity Questionnaire (IPAQ) which is a questionnaire to assess the level of physical activity. This questionnaire obtains the subject's Metabolic Equivalent of Task (MET) of the last week adding up the MET values of the different types of physical activities the subject has done in the last week. Higher values represent a higher level of physical activity.
Changes in emotional eating estimated by the Dutch Eating Behaviour Questionnaire (DEBQ) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in emotional eating will be estimated by the Dutch Eating Behaviour Questionnaire (DEBQ) which is a questionnaire that comprises three scales that measure emotional, external and restrained eating; being 0 the minimum score and 52 the maximum score of the emotional eating scale, 0 the minimum score and 40 the maximum score of the external eating scale and 0 the minimum score and 40 the maximum score of the restrained eating scale. Higher values represent a higher emotional, external or restrained eating.
Changes in the quality of life estimated by the Impact of Weight in the Quality of Life-Lite Questionnaire (IWQOL-Lite) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in the quality of life will be estimated by the Impact of Weight in the Quality of Life-Lite Questionnaire (IWQOL-Lite) which is a questionnaire to assess quality of life in obesity. It comprises five subscales that measure weight-related concerns across five domains: Physical Function, Self-Esteem, Sexual Life, Public Distress and Work. The minimum score of the total punctuation is 31 and the maximum punctuation is 155; the minimum score of the Physical Function scale is 11 and the maximum score is 55; the minimum score of the Self-Esteem scale is 7 and the maximum score is 35; the minimum score of the Sexual Life scale is 4 and the maximum score is 20; the minimum score of the Public Distress scale is 5 and the maximum score is 25 and the minimum score of the Work scale is 4 and the maximum is 20. Higher values represent a higher impact of weight in the quality of life of the individual, in the total score and in each of the domains assessed.
Changes in weight self-stigma estimated by the Weight Self-Stigma Questionnaire (WSSQ) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in weight self-stigma will be estimated by the Weight Self-Stigma Questionnaire (WSSQ) which is a questionnaire to assess weight-related self-stigma that comprises two subscales apart from the total punctuation: self-devaluation and fear of enacted stigma. The minimum score of the total punctuation is 0 and the maximum is 72; the minimum score of the Self-Devaluation subscale is 0 and the maximum is 36; the minimum score of the Fear of Enacted-Stigma subscale is 0 and the maximum is 36. Higher values represent a higher weight-related self-stigma, in the total score and in each of the subscales.

SECONDARY OUTCOMES:
Changes in fat percentage measured by Bio-electrical Impedance Analysis (TANITA) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in fat percentage will be measured by Bio-electrical Impedance Analysis (TANITA).
Changes in muscle mass percentage measured by Bio-electrical Impedance Analysis (TANITA) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in muscle mass percentage will be measured by Bio-electrical Impedance Analysis (TANITA).
Changes in insulin sensitivity measured by homeostasis model assessment (HOMA) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in insulin sensitivity will be measured by homeostasis model assessment (HOMA).
Changes in serum lipid profile | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in total, LDL- and HDL-cholesterol will be measured.
Changes in glucose profile measured by a spectrophotometry | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in the glucose level will be measured by a spectrophotometry.
Changes in waist circumference measured by an inelastic tape (Holtain) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in waist circumference will be measured by an inelastic tape (Holtain).
Changes in blood pressure measured by a sphygmomanometer | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in blood pressure will be measured by a sphygmomanometer.
Changes in general health estimated by the General Health Questionnaire-28 (GHQ-28) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in general health will be estimated by the General Health Questionnaire-28 (GHQ-28), which is a questionnaire to assess the current general health state. Apart from the total punctuation, it comprises four subscales: Somatic Symptoms, Anxiety/Insomnia, Social Dysfunction and Severe Depression. There are two methods to score the GHQ-28. It can be scored from 0 to 3 for each response with a total possible score on the ranging from 0 to 84. Using this method, a total score of 23/24 is the threshold for the presence of distress. Alternatively, the GHQ-28 can be scored with a binary method where "Not at all", and "No more than usual" score 0, and "Rather more than usual" and "Much more than usual" score 1. Using this method, any score above 4 indicates the presence of distress or 'caseness'.
Changes in eating attitudes estimated by the Eating Attitudes Test-12 (EAT-12) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in eating attitudes will be estimated by the Eating Attitudes Test-12 (EAT-12), which is a screening questionnaire to capture undifferentiated eating disorders. Apart from the total punctuation, it comprises three scales: Dieting, Bulimia and food preoccupation and Oral control. The minimum score of the total punctuation is 0 and the maximum score is 36; the minimum score of the Dieting scale is 0 and the maximum score is 12; the minimum score of the Bulimia and food preoccupation is 0 and the maximum score is 12 and the minimum score of the Oral control scale is 0 and the maximum score is 12. Higher values represent further eating problems.
Changes in body image's self-perception estimated by the Figure Rating Scale (FRS) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in body image's self-perception will be estimated by the Figure Rating Scale (FRS), which determines body dissatisfaction in women and men. It consists of nine figures of increasing size with accompanying numerical ratings from 1 to 9. Subjects have to choose two figures that represent how they think they look like and their ideal figure. The higher the discrepancy between these figures, the more subjective body dissatisfaction the individual will have.

OTHER OUTCOMES:
Changes in experiential avoidance estimated by the Acceptance and Action Questionnaire-II (AAQ-II) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in experiential avoidance will be estimated by the Acceptance and Action Questionnaire-II (AAQ-II), which is a questionnaire to assess general experiential avoidance and psychological inflexibility, 7 being the minimum total score and 49 being the maximum total score. Higher values represent higher unwillingness to experience unwanted emotions and thoughts.
Changes in self-compassion level estimated by the Self-Compassion Scale (SCS) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in self-compassion level will be estimated by the Self-Compassion Scale (SCS), which captures this way of being kind and understanding towards oneself in moments of turmoil. Apart from the total punctuation (overall self-compassion), it comprises six subscales that assess components of self-compassion across three related facets: Self-Kindness/Self-Judgment, Common Humanity/Isolation and Mindfulness/Over-Identification. The minimum total score is 12 and the maximum total score is 60; the minimum score of the Self-Kindness/Self-Judgment subscale is 4 and the maximum score is 20; the minimum score of the Common Humanity/Isolation subscale is 4 and the maximum score is 20; the minimum score of the Mindfulness/Over-Identification scale is 4 and the maximum score is 20. Higher values represent higher overall self-compassion.
Changes in mindfulness abilities measured by the Five Facets Mindfulness Questionnaire (FFMQ) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in mindfulness abilities will be measured by the Five Facets Mindfulness Questionnaire (FFMQ), which is a questionnaire to assess the ability of mindfulness of the individual. Apart from the total punctuation, it comprises five subscales referring to five facets of mindfulness: Observe, Describe, Act with Awareness, Nonjudge of Inner Experience and Non-React to Inner Experience. The minimum score of the total punctuation is 39 and the maximum score is 195; the minimum score of the Observe subscale is 8 and the maximum score is 40; the minimum score of the Describe subscale is 8 and the maximum score is 40; the minimum score of the Act with Awareness subscale is 8 and the maximum score is 40; the minimum score of the Nonjudge of Inner Experience subscale is 8 and the maximum score is 40 and the minimum score of the Non-React to Inner Experience subscale is 7 and the maximum score is 35.
Changes in avoidance and inflexibility in relation to difficult weight-related thoughts and feelings estimated by the Acceptance and Action Questionnaire for Weight-Related Problems (AAQ-W) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in avoidance and inflexibility in relation to difficult weight-related thoughts and feelings will be estimated by the Acceptance and Action Questionnaire for Weight-Related Problems (AAQ-W), which is a questionnaire to assess the acceptance of weight-related feelings, defusion from weight related thoughts, and the degree to which thoughts and feelings interfere with valued action, 22 being the minimum score and 154 being the maximum score of the total punctuation. Higher values represent higher experiential avoidance and psychological inflexibility in relation to difficult weight-related thoughts and feelings.
Changes in body image flexibility estimated by the Body Image-Acceptance and Action Questionnaire (BI-AAQ) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in body image flexibility will be estimated by the Body Image-Acceptance and Action Questionnaire (BI-AAQ), which is a questionnaire to assess body image flexibility, 12 being the minimum total score and 84 being the maximum total score. Higher values represent higher body image flexibility.
Changes in the fit between participant's actual activities and the valued behavioral pattern measured by Valued Living Questionnaire (VLQ) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in the fit between participant's actual activities and the valued behavioral pattern will be measured by Valued Living Questionnaire (VLQ), which is a two part instrument to assess valued living. In the first part, subjects rate the importance of 10 domains of living on a 10 point Likert style scale (1 being "not at all important" and 10 being "extremely important") and the second part consists on rating, using a 10 point Likert style scale, how consistently he or she has lived in accord with the valued behavioral pattern within each domain over the past week (1 being "not at all consistent" and 10 being "extremely consistent"). Higher values in the second part represent higher fit between the subject's actual activities and the valued behavioral pattern.
Changes in cognitive fusion measured by the Cognitive Fusion Questionnaire (CFQ) | Pretreatment-Posttreatment (5 months)-7 months follow-up
  Changes in cognitive fusion will be measured by the Cognitive Fusion Questionnaire (CFQ), which is a questionnaire to assess the extent to which an individual is psychologically tangled with and dominated by the form or content of his or her thoughts, 7 being the minimum total score and 49 being the maximum total score. Higher values represent higher cognitive fusion.

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Maiz Aldalur, PhD, Principal Investigator — Assistant teacher in the Department of Personality, Assessment and Psychological Treatments of the Faculty of Psychology of the Basque Country University (EHU/UPV); Enrique Echeburúa Odriozola, Professor, Principal Investigator — Professor in Clinical Psychology in the Department of Personality, Assessment and Psychological Treatments of the Faculty of Psychology of the Basque Country University (EHU/UPV)
Locations (1):
- Department of Personality Assesment and Psychological Treatments of the Faculty of Psychology of the Basque Country University (UPV/EHU), Donostia / San Sebastian, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iturbe I, Pereda-Pereda E, Echeburua E, Maiz E. The Effectiveness of an Acceptance and Commitment Therapy and Mindfulness Group Intervention for Enhancing the Psychological and Physical Well-Being of Adults with Overweight or Obesity Seeking Treatment: The Mind&Life Randomized Control Trial Study Protocol. Int J Environ Res Public Health. 2021 Apr 21;18(9):4396. doi: 10.3390/ijerph18094396. PMID 33919059